CLINICAL TRIAL: NCT06090240
Title: Maximizing Teachable Moments: Motivational Interviewing (MI) to Enhance Advance Care Planning (ACP) for Older Adults and Caregivers After Emergency Visits - A Mixed-Method Randomized Controlled Trial
Brief Title: Motivational Interviewing to Enhance Advance Care Planning for Older Adults and Caregivers After Emergency Visits
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-2023-150, HKWC-2023-342
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Older Adults; Advance Care Planning; Advance Directives; Family Members

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interview (Experimental): Older adult-family member dyads in this arm will receive an MI-based education intervention our team developed.
  Interventions: Other: MI-based ACP intervention
- Self-learning (No Intervention): Older adult-family member dyads in this arm will receive a self-learning ACP educational material developed by the Hong Kong Hospital Authority.

INTERVENTIONS:
Other: MI-based ACP intervention — Motivational Interviewing on Advance Care Planning Intervention: Dyads of older adults and family caregivers will receive three MI-based ACP counselling sessions: (1) a preparatory session, (2) motivation session, and (3) planning session. The preparatory session will take 10-15 minutes, and the following two sessions in weeks 2 and 3 will last 30-45 minutes each. Before each session, the nurse interventionist will first assess the dyad's readiness to engage in ACP based on the state of change algorithm. Participants who have never thought about ACP will be in the pre-contemplation state, those who are willing to discuss EOL care and preferences to be in the contemplation state, those ready to talk about EOL planning to be in the preparation state, and those in the action state have a confirmed action plan on signing up their ADs. Readiness-based ACP goals will be established, and state-matched MI counseling will be customized for each participant.
  Arms: Motivational Interview

SUMMARY:
This study aims to evaluate the effectiveness of a motivational interviewing (MI) intervention in enhancing advance care planning (ACP) among older adults who have visited the Emergency Room (ER) in the past six months and their family caregivers. The main question it aims to answer is: The effectiveness of the MI-based ACP intervention implemented within six months of an ER visit on improving older adults' advance directives (AD) completion rate.

Compared to participants in the control group who will only receive a self-education booklet, participants in the intervention group will receive a motivational interview educational intervention to see the effectiveness of an MI-based ACP intervention implemented within six months following an emergency room visit regarding the completion of AD for older adults.

DETAILED DESCRIPTION:
Targeted issue: At present no feasible method exists to empower older adults following ER visits to engage in ACP in Hong Kong.

Population: The target group will be dyads comprising older adults who have had ER visits within the previous six months and their family caregivers.

Intervention: An MI-based ACP intervention our team developed.

Main study aim: To investigate the effectiveness of an MI-based ACP intervention implemented within six months following an emergency room visit on completion of AD for older adults compared to a self-education group.

Study method: Investigators will recruit eligible participants from two largest public hospitals, including the geriatric outpatient clinic of Queen Mary Hospital (IRB Ref: UW23-402) and the accident & emergency department of Queen Elizabeth Hospital (IRB Ref: KC/KE-23-0058/ER-1). A parallel RCT (allocation ratio= 1:1) with a post-trial qualitative study will be adopted and three follow-up time points at 3-, 6- and 12-month post-intervention. Participants in the intervention group will receive a motivational interview educational intervention, while participants in the comparison group will receive the pictorial ACP educational booklet for self-learning only. Completion of AD and health service utilization will be assessed at three follow-up time points. In addition, a post-intervention interview, regarding stakeholders' views on the relevance, effectiveness, and experience of the intervention., will be conducted.

ELIGIBILITY:
The target group will be dyads comprising older adults who have had ER visits within the previous six months and their family caregivers. A dyad is defined as one older adult and one primary family caregiver of the older adult.

For older adults:

Inclusion Criteria:

* Aged 65 or older
* At least one episode of ER visit in the last six months
* Has a family caregiver to be present during the intervention
* Able to communicate in Chinese

Exclusion Criteria:

* Has completion of an AD
* Moderate to severe cognitive impairment or diagnosis of dementia, as identified in health records
* Communication problems (e.g., deafness or aphasia)

For family caregivers:

Inclusion Criteria:

* Aged 18 or above
* Immediate or extended family member or friend nominated by an eligible older adult participant as primary caregiver
* Able to communicate in Chinese

Exclusion Criteria:

* Moderate to severe cognitive impairment
* Communication problems (e.g., deafness or aphasia)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Older adults' readiness for ACP | before the intervention (T0), and 3-month (T1), 6-month (T2), and 12-months (T3) post intervention.
  Older adults' readiness for ACP (primary outcome) will be measured by the readiness subscales of the Advance Care Planning Engagement Survey (ACPES), which comprises 6 items rated on a 5-point Likert scale, ranging from 1 (worst outcome) to 5 (best outcome). A higher score indicates a higher readiness for ACP. It assesses an individual's readiness to sign official papers for health decision delegates and ADs and readiness to talk with family and physicians about EOL care, and has been validated in Hong Kong.

SECONDARY OUTCOMES:
Family caregivers' readiness for ACP | before the intervention (T0), and 3-month (T1), 6-month (T2), and 12-months (T3) post intervention.
  Family caregivers' readiness for ACP will be measured by the researcher-developed family caregivers' ACP engagement survey (FACP-10), which consists of 10 items rated on a 5-point Likert scale, ranging from 1 (worst outcome) to 5 (best outcome). A Higher score indicates a higher readiness for ACP. The survey assesses family caregivers' self-reported levels of ACP knowledge, readiness to discuss ACP with a loved one, self-efficacy in initiating ACP conversations with a loved one and barriers to such initiation, and emotional perceptions of and attitudes toward ACP, as well as whether having the necessary communication tools for ACP conversations. We developed the instrument based on the key domains reported in ACPES and the constructs identified in a systematic review of family caregivers' roles in ACP. Our pilot data demonstrated adequate reliability of the scale in Hong Kong family caregivers.
Older adults' emotional perception of ACP | before the intervention (T0), and 3-month (T1), 6-month (T2), and 12-months (T3) post intervention.
  Older adults' emotional perception of ACP will be measured by the 3 item self-efficacy subscale (SE-3) of the ACPES on a 5-point Likert scale, ranging from 1 (worst outcome) to 5 (best outcome), with higher scores indicating greater confidence about participating in ACP. The scale has been validated in Chinese.
Older adults' and family caregivers' decisional conflict | before the intervention (T0), and 3-month (T1), 6-month (T2), and 12-months (T3) post intervention.
  Decisional conflict will be measured by both older adults' and family caregivers' responses to the Decisional Conflict Scale (DCS), which consists of 16 items in 5 domains (informed, values clarity, support, uncertainty, and effective decision) scored on a 5-point Likert scale, ranging from 1 (worst outcome) to 5 (best outcome). A Higher scores indicate more decisional conflict when considering goal of EOL care. The DCS has been validated in a Chinese population.
Older adults and family caregivers' congruence in goal of EOL care | before the intervention (T0), and 3-month (T1), 6-month (T2), and 12-months (T3) post intervention.
  Congruence in goal of EOL care will be assessed by the dyad's response to a scenario case (DSC-2) separately "in the event that I (the older adult participant) am in the terminal ill situation …." Each member of the dyad will independently choose one of three options: "the goals of care should be focused on prolonging my (his/her) life, no matter what it may cost," "b. the goals of care should be focused on my (his/her) comfort and peace, even though it may not extend life" or "I am not sure." The responses will be stratified and compared to assess the degree of congruence between older adults and family caregivers.
Older adults' completion of AD documentation | before the intervention (T0), and 3-month (T1), 6-month (T2), and 12-months(T3) post intervention .
  Older adults' completion of AD documentation will be measured by reviewing participants' medical records for a new AD document during the study follow-up period.
Older adults' health service utilization | 3-month (T1), 6-month (T2), and 12-months (T3) post intervention.
  Older adults' health service utilization will be measured by participant self-reports of the number and duration of unplanned ER visits and hospital admissions.
Older adults' and family caregivers' baseline characteristics | before the intervention (T0)
  Older adults' and family caregivers' baseline characteristics will be assessed by a survey on demographics, disease information, previous ACP-related experience, social support, and mental and physical health status.
Older adults and family caregivers' experience with the Nurse Navigation Program | 3-month (T1) post intervention
  The older adults and family caregivers will be interviewed together about their experience and perception of the intervention, the logistics of the intervention, and how it could be improved in the future. The interview questions will include: 1) What was your overall feeling about the NNP? 2) Tell me your opinion of the NNP's impact on your ACP decision-making. 3) Which parts of the NNP were the most or least helpful? 4) How did you benefit from participating in the NNP? 5) What are the NNP's limitations? 6) What changes need to be made to render the NNP more helpful for future participants?

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Chin LIN, PhD,FAAN,RN, Principal Investigator — University of Hong Kong, School of Nursing
Locations (1):
- University of Hong Kong, School of Nursing, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No